CLINICAL TRIAL: NCT05190003
Title: Effect of Supervised, Short-term Stabilization Exercises on the Pain, Posture Control, Balance, Functional Tests and Pressure Distribution in Patients After First-time, Single-level Lumbar Spine Microdiscectomy.
Brief Title: Influence of Supervised Stabilization Exercises on Postural Control in Patients After Spine Surgery.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Gdansk University of Physical Education and Sport (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DZN/1/2021/PP
Record Dates: First submitted 2021-11-19; First posted 2022-01-13 (Actual); Last update posted 2022-09-13 (Actual); Status verified 2022-09

CONDITIONS: Low Back Pain
Keywords: Low back pain,; Microdiscectomy,; Lumbar disc herniation,; Functional exercise,; Lumbar Stabilization Exercise
MeSH Terms: conditions — Low Back Pain; Intervertebral Disc Displacement | interventions — Non-Randomized Controlled Trials as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group I: The first time of patients attending single-level lumbar microdiscectomy (Experimental): Study group I:
  On the basis of neurosurgical examination and MRI imaging, 40 patients aged 20-65 years with pains in the lumbar spine will be referred for the first-time single-level microdiscectomy procedure. Microdiscectomy patients will begin a rehabilitation program that will be includes exercises to reduce pain and strengthen the stabilizing muscles of the lumbar spine. From week to week, exercises will be difficult, among others due to the change of initial positions, the number of repetitions of exercises, or a longer duration of isometric exercises.
  Interventions: Other: Experimental Study
- Study group II: Control healthy people (No Intervention): Study group II:
  40 people aged 20-65 years. Including criteria: healthy persons without lumbar spine pain for at least 6 months and without lumbar spine surgery.

INTERVENTIONS:
Other: Experimental Study — On the basis of neurosurgical examination and MRI imaging, 40 patients aged 20-65 years with pains in the lumbar spine will be referred for the first-time single-level microdiscectomy procedure. Microdiscectomy patients will begin a rehabilitation program that will be includes exercises to reduce pain and strengthen the stabilizing muscles of the lumbar spine. From week to week, exercises will be difficult, among others due to the change of initial positions, the number of repetitions of exercises, or a longer duration of isometric exercises.
  Arms: Study group I: The first time of patients attending single-level lumbar microdiscectomy

SUMMARY:
The aim of the study is to determine the impact of early rehabilitation in patients after lumbar spine surgery using microdiscectomy on balance, postural stability and foot pressure distribution. The tests will be carried out at the Physical Effort Laboratory in Gdańsk.

DETAILED DESCRIPTION:
Back pain (LBP) has become a major public health problem. In the case of pain in the lumbar spine, conservative or surgical treatment is used. In conservative treatment, patients undergo an appropriate rehabilitation program or use painkillers / anti-inflammatory drugs. When conservative treatment is unsuccessful, patients based on the MRI image and neurosurgical consultation are referred to the lumbar spine microdiscectomy. Therefore, patients consciously and voluntarily can start research on the effect of supervised exercises to stabilize the lumbar spine after single-level lumbar spine microdiscectomy on pain reduction, pressure distribution, balance, posture control, and basic functional tests.

Before the operation, during the first examinations, patients are informed about the ergonomic and behavioral procedure after the operation, and rehabilitation program. After surgery, a supervised exercise program begins three times a week for a month, lead by a qualified physiotherapist. Supervision is carried out online using generally available applications, including WhatsApp, messenger. After one month, patients are re-examined in the same way as before the surgery. The rehabilitation program after the microdiscectomy of the lumbar spine enables the voluntary extension of rehabilitation for another two months. During subsequent meetings with a physiotherapist, patients are taught new exercises that differ from week to week in terms of difficulty in performing, the number of repetitions, and the time to maintain tension.

Moreover, in the third month of the rehabilitation program, exercises with the use of a sensorimotor disc are planned. After completing the rehabilitation program, patients are invited for follow-up examinations six months and one year after the end of rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* age 20 to 65 years, neurosurgical assessment and MRI imagine,discopathy, pernament low back pain with or without radiating to the lower limb.

Exclusion Criteria:

* patients beyond the age range, a previous lumbar spinal operation, spinal tumors, new fractures, intolerance of rehabilitation programs.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-10 (Actual); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
Modified Schober's Test | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  The test is used to assess the flexibility, active range of motion of the lumbar spine. During the examination, the patient assumes a standing position, and the examiner marks a point at the level of the intervertebral space L₅ - S₁. Then he marks the points: 10 cm above and 5 cm below. The examined person is asked to bend the torso as far as possible, the examiner measures the difference in distance from the marked points.
Chair Stand Test (CST) | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  The test is used to assess the ability to stand up and down on a chair and lower body strength. The patient is asked to stand up to an upright position and sit with his arms crossed over his chest from a chair of standard height (43 cm) as many times as he can within 30 seconds. Blood pressure and heart rate measurements are collected before and after the test.
"Timed Get-up-and-Go" Test | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  This test determines fall risk and measures the progress of balance, sit to stand, and walking. During the test, the patient must get up from the chair and walk 3 meters as quickly as possible and sit down again. A patient has two trials. The better sample is analyzed.

SECONDARY OUTCOMES:
Body Mass Index (BMI) | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  Each participant's weight and height will be assessed to determine their BMI using the formula weight [kg] / height [m] 2. This will be interpreted in line with the international cut-off points. In addition, body composition will be analyzed using bioelectric impedance.
Fingertip-to-Floor Test | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  During the test, the subject keeps the feet connected and does not lift them. The patient is asked to bend his torso forward by reaching with his fingertips to the ground with straightened knees, elbows and toes. The examiner measures the vertical distance between the tip of the middle finger and the ground.
Romberg's Trial | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  During the test, the subject keeps the feet connected and does not lift them. The patient is asked to bend his torso forward by reaching with his fingertips to the ground with straightened knees, elbows and toes. The examiner measures the vertical distance between the tip of the middle finger and the ground.
Tandem Romberg Test | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  Tandem Romberg test (tandem stance without shoes and eyes closed) with a non-dominant foot in front of the dominant one. The arms hang down along the body. The examiner measures the time in seconds with a stopwatch. During the test, the test is interrupted when the patient tears off his feet, opens his eyes, touches the wall with his hand / arm. The test is performed three times and the arithmetic mean of these results is calculated.
Biodex Balance System SD | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  The study will carry out three tests: a postural stability test on a stable platform, a dynamic test for assessing risk of fall using a difficulty level of 12 to 8, and a difficulty level of 8. During the test patient is asked to keep the market as close as possible to the center of the target appearing on the monitor screen. The patient's score in this test depends on the number of deviations from the center, therefore the lower the score the better.
  It will be performed during three attempts of 20 seconds each. The system calculates the mean of the three trials. The examine's person stands on a static platform without shoes and feet are placed freely. Three indicators are obtained: the Overall Postural Stability Index (OSI), the Anterior / Posterior Postural Stability Index (AP) and the Medial / Lateral Postural Stability Index (ML). The tests are performed with eyes open and closed.
Visual Analogue Scale (VAS) | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  The level of pain in the lumbar spine and lower extremities after microdiscectomy, it's assessed on the basis of the visual analog scale (VAS); A 10 cm scale where 0 means "no pain" and 10 "the worst pain imaginable.
Oswestry Low Back Pain Disability Questionnaire (ODI) | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  The Oswestry Disability Index (ODI) is a tool that assesses the level of disability of patients with back pain syndromes and the associated limitations in functioning in various spheres of life. ODI consists of 10 sections.The total score is multiplied by 2 and expressed as a percentage. The result in the range of 0-20% indicates a minimum level of disability, while 81-100% indicates a significant disability.
Spine Tango Questionnaire | T1-pre-intervention,T2-after first month the intervention,T3-after second month the intervention, T4-after third month the intervention, T5- after six months the intervention, T6-after twelve months the intervention.
  The questionnaire, which includes questions, among others of pain intensity level measured separately on graphic scales of 0-10 ratings, overall quality of life, social disability and incapacity for work - each on a five-point scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Gdansk University of Physical Education and Sport, Gdansk, Poland